CLINICAL TRIAL: NCT03259087
Title: A 2-Part, Open-Label Trial to Evaluate the Pharmacokinetics of MK-3866 Following the Administration of a Single IV Dose to Subjects With Mild, Moderate, and Severe Renal Impairment and End Stage Renal Disease
Brief Title: Pharmacokinetics (PK) and Safety of a Single Intravenous (IV) Dose of MK-3866 in Participants With Impaired Renal Function and in Healthy Controls (MK-3866-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3866-005; CA22640 (Other: Celerion); MK-3866-005 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Mild Renal Impairment (Experimental): Participants receive a single IV infusion of 200 mg MK-3866 over 30 minutes on Day 1.
  Interventions: Drug: MK-3866
- Part 1: Moderate Renal Impairment (Experimental): Participants receive a single IV infusion of 200 mg MK-3866 over 30 minutes on Day 1.
  Interventions: Drug: MK-3866
- Part 1: Severe Renal Impairment (Experimental): Participants receive a single IV infusion of 200 mg MK-3866 over 30 minutes on Day 1.
  Interventions: Drug: MK-3866
- Part 1: Healthy Participants (Experimental): Participants receive a single IV infusion of 200 mg MK-3866 over 30 minutes on Day 1.
  Interventions: Drug: MK-3866
- Part 2: End-stage Renal Disease Undergoing Hemodialysis (Experimental): End-stage renal disease (ESRD) participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1 just after hemodialysis (HD) in Period 1 and just before HD in Period 2. There was a washout of at least 6 days before dosing in Period 2.
  Interventions: Drug: MK-3866

INTERVENTIONS:
Drug: MK-3866 — Single IV infusion of 200 mg administered over 30 minutes (±5 minutes) on Day 1 of each treatment period.

SUMMARY:
The purpose of this study is to compare plasma and urine PK parameters of MK-3866 between participants with impaired renal function and healthy control participants, to investigate the extent to which MK-3866 is removed from the plasma by hemodialysis (HD), and evaluate the safety and tolerability of MK-3866 in participants with impaired renal function.

DETAILED DESCRIPTION:
This is an open-label, 2-part single dose study: Part 1 will include participants with mild, moderate, and severe renal impairment (as well as healthy control participants), and Part 2 will include participants with end stage renal disease (ESRD) undergoing HD. Participants in Part 1 will receive a single IV dose of MK-3866, and plasma and urine samples will be collected over pre-specified time intervals. Participants in Part 2 will receive a single IV dose of MK-3866 on two separate occasions: in Period 1 immediately following their normally-scheduled HD, and in Period 2 approximately 30 minutes prior to their normally-scheduled HD. Plasma, urine, and dialysate samples will be collected over pre-specified time intervals for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential. Male participants with female partner(s) of child-bearing potential agree to use a medically acceptable method of contraception during the study and for 90 days after dosing. If partner is pregnant, males agree to use a condom; if partner is of child-bearing potential, partner must use additional birth control
* Male participants agree not to donate sperm from the first dose until 90 days after dosing
* Adequate venous access

Renal Impaired Participants

* Liver function tests (serum alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) and serum bilirubin (total and direct) within upper limit of normal
* Panels A, B, and C: no clinically significant change in renal status at least 1 month prior to dosing and not currently or previously been on hemodialysis
* Panel E only: ESRD maintained on stable regimen of at least 3 times per week HD for at least 3 months prior to first dosing

Healthy Participants

* Age within ± 15 years of the mean age of participants with impaired renal function to which the healthy participant is matched
* Medically healthy as per medical history, physical examination, vital signs, 12-lead electrocardiograms (ECGs), and clinical laboratory safety tests
* Blood urea nitrogen, liver function tests (ALT, AST, alkaline phosphatase [ALP]), and serum bilirubin (total and direct) within upper limit of normal.

Exclusion Criteria:

* Mentally/legally incapacitated, or significant emotional problems or significant psychiatric disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, respiratory, genitourinary or major neurological abnormalities or diseases
* History of any illness that might confound the results of the study or poses an additional risk to the participant by their participation in the study
* Clinically significant history of cancer
* Smoker and/or has used nicotine or nicotine-containing products within 3 months prior to screening
* Female participants of childbearing potential, pregnant, or lactating
* Positive results for urine or saliva drug screen and/or urine or breath alcohol screen at screening or check-in
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)
* Consumes more than 3 glasses of alcoholic beverages within 6 months of screening
* Consumes excessive amounts of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day
* Major surgery, donated or lost 1 unit of blood within 4 weeks prior to screening, or donated plasma within 7 days prior to dosing in Part 1 or first dose in Part 2

Renal Impaired Participants

* Panels A, B, and C: Failed renal transplant or has had nephrectomy
* Panels A, B, and C: Rapidly fluctuating renal function, as determined by historical measurements; or demonstrated/suspected renal artery stenosis
* Panel E only: Has required frequent emergent HD (≥3) within a year prior to first dosing

Healthy Participants

* Renal transplant or nephrectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami ( Site 0001), Hialeah, Florida
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Mild Renal Impairment (RI): Participants received a single intravenous (IV) infusion of MK-3886 200 mg over 30 minutes on Day 1.
- Part 1: Moderate Renal Impairment; Part 1: Severe Renal Impairment; Part 1: Healthy Participants: Participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1.
Period: Part 1 and Period 1 of Part 2
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 1: Healthy Participants | Part 2: End-stage Renal Disease Undergoing Hemodialysis
Started | 8 | 8 | 8 | 10 | 8
Completed | 8 | 8 | 8 | 10 | 7
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Period 2 of Part 2
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 1: Healthy Participants | Part 2: End-stage Renal Disease Undergoing Hemodialysis
Started | 0 (Period 2 did not apply to Part 1 participants) | 0 (Period 2 did not apply to Part 1 participants) | 0 (Period 2 did not apply to Part 1 participants) | 0 (Period 2 did not apply to Part 1 participants) | 7
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 1: Healthy Participants | Part 2: End-stage Renal Disease Undergoing Hemodialysis | Total
Number analyzed (Participants) | 8 | 8 | 8 | 10 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (5.65) | 67.0 (9.24) | 57.3 (13.83) | 61.2 (8.36) | 51.9 (8.68) | 61.1 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 4 | 3 | 15
  Male | 4 | 6 | 6 | 6 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 4 | 1 | 15
  Not Hispanic or Latino | 6 | 4 | 4 | 6 | 7 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 7 | 15
  White | 6 | 6 | 5 | 8 | 1 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28.125 [20.00 to 36.00] | 27.625 [23.00 to 34.00] | 28.625 [20.00 to 32.00] | 28.800 [27.00 to 30.00] | 29.875 [27.00 to 34.00] | 28.619 [20.00 to 36.00]

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve of MK-3866 From Time Zero to Infinity (AUC0-inf)
Description: Plasma samples were collected at pre-specified time points and AUC0-inf was assessed. Plasma concentrations of MK-3866 were determined using high-performance liquid chromatography with tandem mass spectrometry (HPLC-MS/MS).
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 36, and 48 hours after dosing on Day 1, and 60 and 72 hours after dosing for Severe Renal Impairment participants
Population: All participants who received MK-3866 infusion. Healthy participants were those who matched gender, and mean age and BMI of the comparator experimental group(s).
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Groups:
- Part 1: Healthy Participants (Mild + Moderate RI): Participants received a single intravenous (IV) infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender and mean age and BMI of the combined mild and moderate RI groups
- Part 1: Healthy Participants (Severe RI): Participants received a single intravenous (IV) infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender and mean age and BMI of the severe RI group.
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
µM*hr | 104 [87.2 to 125] | 141 [115 to 174] | 83.5 [75.0 to 92.9] | 244 [169 to 352] | 81.8 [72.4 to 92.4]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.25, 90% CI 2-sided [1.07 to 1.47] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.70, 90% CI 2-sided [1.42 to 2.02] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 2.98, 90% CI 2-sided [2.20 to 4.04] — GMR is ratio of Experimental Group / Healthy Group

2. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve of MK-3866 From Time Zero to the Time of the Last Quantifiable Sample (AUC0-last)
Description: Plasma samples were collected at pre-specified time points and AUC0-last was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
µM*hr | 103 [86.7 to 123] | 139 [114 to 170] | 83.0 [74.5 to 92.5] | 237 [166 to 338] | 81.4 [72.0 to 92.0]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.25, 90% CI 2-sided [1.06 to 1.46] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.68, 90% CI 2-sided [1.41 to 1.99] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 2.91, 90% CI 2-sided [2.17 to 3.90] — GMR is ratio of Experimental Group / Healthy Group

3. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve of MK-3866 From Time Zero to 24 Hours After Dosing (AUC0-24)
Description: Plasma samples were collected at pre-specified time points and AUC0-24 was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, and 24 hours after dosing on Day 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
µM*hr | 96.2 [82.0 to 113] | 127 [107 to 152] | 79.7 [71.6 to 88.7] | 182 [136 to 243] | 78.1 [69.2 to 88.3]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.21, 90% CI 2-sided [1.04 to 1.40] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.59, 90% CI 2-sided [1.36 to 1.86] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 2.32, 90% CI 2-sided [1.82 to 2.97] — GMR is ratio of Experimental Group / Healthy Group

4. Primary Outcome: Part 1: Plasma Concentration of MK-3866 at the End of the Infusion (Ceoi)
Description: Plasma samples were collected at pre-specified time points and Ceoi was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: At the end of the infusion (0.5 hours after infusion start) on Day 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
µM | 26.6 [22.3 to 31.8] | 27.7 [24.2 to 31.7] | 27.0 [23.9 to 30.5] | 29.7 [25.4 to 34.7] | 26.9 [23.7 to 30.5]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.99, 90% CI 2-sided [0.84 to 1.16] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.03, 90% CI 2-sided [0.90 to 1.18] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.11, 90% CI 2-sided [0.95 to 1.29] — GMR is ratio of Experimental Group / Healthy Group

5. Primary Outcome: Part 1: Maximum Plasma Concentration of MK-3866 (Cmax)
Description: Plasma samples were collected at pre-specified time points and Cmax was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: as for outcome 1
Population: All participants who received MK-3866 infusion. Healthy participants were those who matched gender, and mean age and BMI of the combined comparator experimental groups.
Measure: Mean (95% Confidence Interval); unit: µM
Groups:
- Part 1: Healthy Participants (Mild, Moderate, and Severe RI): Participants received a single intravenous (IV) infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender and mean age and BMI of the mild, moderate, and severe groups.
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Mild, Moderate, and Severe RI)
Number analyzed (Participants) | 8 | 8 | 8 | 10
µM | 27.4 [26.0 to 28.9] | 28.0 [26.4 to 29.7] | 28.7 [26.4 to 31.2] | 26.7 [24.8 to 28.8]

6. Primary Outcome: Part 1: Plasma Clearance of MK-3866 (CL)
Description: Plasma samples were collected at pre-specified time points and CL was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
L/hr | 3.80 [3.17 to 4.55] | 2.80 [2.28 to 3.44] | 4.75 [4.27 to 5.28] | 1.62 [1.12 to 2.35] | 4.85 [4.29 to 5.48]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.80, 90% CI 2-sided [0.68 to 0.94] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.59, 90% CI 2-sided [0.49 to 0.70] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.34, 90% CI 2-sided [0.25 to 0.45] — GMR is ratio of Experimental Group / Healthy Group

7. Primary Outcome: Part 1: Time to Maximum Plasma Concentration of MK-3866 (Tmax)
Description: Plasma samples were collected at pre-specified time points and Tmax was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
Hours | 0.50 [0.47 to 0.50] | 0.49 [0.47 to 0.50] | 0.50 [0.47 to 0.50] | 0.50 [0.47 to 0.53] | 0.50 [0.47 to 0.50]

8. Primary Outcome: Part 1: Elimination Terminal Half-life of Plasma MK-3866 (t1/2)
Description: Plasma samples were collected at pre-specified time points and t1/2 was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric % coefficient of variation (%CV).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
Hours | 7.38 (13.3) | 8.23 (17.0) | 7.00 (12.7) | 14.7 (17.8) | 6.90 (13.0)

9. Primary Outcome: Part 1: Volume of Distribution of Plasma MK-3866 (Vz)
Description: Plasma samples were collected at pre-specified time points and Vz was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
Liters | 40.4 (18.3) | 33.3 (18.0) | 48.0 (17.3) | 34.4 (29.5) | 48.3 (17.7)

10. Primary Outcome: Part 2: AUC0-inf of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and AUC0-inf was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, 24, 36, 48, 60, and 72 hours after dosing on Day 1 of Period 1 and 2, and 2.5, 3.5, and 4 hours after dosing on Day 1 of Period 2
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Groups:
- Part 2, Period 1: ESRD Undergoing HD (Dosed After HD): Participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1 just after HD in Period 1. There was a washout of at least 6 days before dosing in Period 2.
- Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD): Participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1 just before HD in Period 2. There was a washout of at least 6 days before dosing in Period 2.
- Part 1: Healthy Participants (ESRD): Participants received a single intravenous (IV) infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender and mean age and BMI of the ESRD group.
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
µM*hr | 323 [260 to 401] | 129 [103 to 161] | 81.3 [70.6 to 93.7]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 3.97, 90% CI 2-sided [3.26 to 4.82] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.58, 90% CI 2-sided [1.30 to 1.92] — GMR is ratio of Experimental Group / Healthy Group

11. Primary Outcome: Part 2: AUC0-last of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and AUC0-last was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
µM*hr | 294 [241 to 358] | 118 [97.4 to 144] | 80.9 [70.2 to 93.3]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 3.63, 90% CI 2-sided [3.03 to 4.36] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.46, 90% CI 2-sided [1.22 to 1.75] — GMR is ratio of Experimental Group / Healthy Group

12. Primary Outcome: Part 2: AUC0-24 of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and AUC0-24 was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 3, 4.5, 6, 8, 10, 12, and 24 hours after dosing on Day 1 of Period 1 and 2, and 2.5, 3.5, and 4 hours after dosing on Day 1 of Period 2
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
µM*hr | 203 [174 to 238] | 84.7 [74.6 to 96.1] | 77.8 [67.5 to 89.6]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 2.61, 90% CI 2-sided [2.23 to 3.06] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 1.09, 90% CI 2-sided [0.95 to 1.25] — GMR is ratio of Experimental Group / Healthy Group

13. Primary Outcome: Part 2: Ceoi of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and Ceoi was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: At the end of the infusion (0.5 hours after infusion start) on Day 1 of Period 1 and Period 2
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
µM | 26.3 [22.7 to 30.3] | 25.3 [19.1 to 33.4] | 26.8 [23.1 to 31.0]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.98, 90% CI 2-sided [0.84 to 1.14] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.94, 90% CI 2-sided [0.75 to 1.20] — GMR is ratio of Experimental Group / Healthy Group

14. Primary Outcome: Part 2: Cmax of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and Cmax was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
µM | 26.6 [23.1 to 30.6] | 25.3 [19.1 to 33.4] | 26.8 [23.1 to 31.0]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.99, 90% CI 2-sided [0.85 to 1.16] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.94, 90% CI 2-sided [0.75 to 1.20] — GMR is ratio of Experimental Group / Healthy Group

15. Primary Outcome: Part 2: CL of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and CL was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
L/hr | 1.23 [0.989 to 1.53] | 3.08 [2.47 to 3.85] | 4.87 [4.23 to 5.61]
Statistical Analysis 1: Comparison: Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.25, 90% CI 2-sided [0.21 to 0.31] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) vs Part 1: Healthy Participants (ESRD); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.63, 95% CI 2-sided [0.52 to 0.77] — GMR is ratio of Experimental Group / Healthy Group

16. Primary Outcome: Part 2: Tmax of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and Tmax was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
Hours | 0.50 [0.50 to 0.75] | 0.50 [0.50 to 0.50] | 0.48 [0.47 to 0.50]

17. Primary Outcome: Part 2: t1/2 of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and t1/2 was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1. Method of dispersion used for these data is geometric %CV.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
Hours | 20.9 (21.6) | 20.0 (18.0) | 6.81 (13.2)

18. Primary Outcome: Part 2: Vz of Plasma MK-3866
Description: Plasma samples were collected at pre-specified time points and Vz was assessed. Plasma concentrations of MK-3866 were determined using HPLC-MS/MS. For ESRD participants, hemodialysis took place predose in Period 1 and from 0.5 to 4.5 hours after dosing in Period 2. Data for healthy participants are from Part 1. Method of dispersion used for these data is geometric %CV.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 8 | 7 | 8
Liters | 37.1 (20.0) | 89.1 (12.2) | 47.9 (18.8)

19. Secondary Outcome: Part 1: Total Amount of MK-3866 Excreted in the Urine Over 24 Hours (Ae0-24)
Description: Urine samples were collected at pre-specified intervals and Ae0-24 was assessed. Ae0-24 was obtained by adding the amounts excreted over each collection interval. Urine concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
mg | 97.1 [79.6 to 118] | 69.2 [48.4 to 98.8] | 107 [89.0 to 130] | 34.6 [22.7 to 52.6] | 115 [96.4 to 137]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.90, 90% CI 2-sided [0.74 to 1.11] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.64, 90% CI 2-sided [0.47 to 0.88] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.30, 90% CI 2-sided [0.21 to 0.43] — GMR is ratio of Experimental Group / Healthy Group

20. Secondary Outcome: Part 1: Renal Clearance (CLr) of MK-3866
Description: Urine samples were collected at pre-specified intervals and CLr was assessed. CLr was calculated as AE(t'-t")/AUC(t'-t"), where t'-t" is the longest interval of time during which AE and AUC are both obtained. Urine concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
L/hr | 2.00 [1.50 to 2.66] | 1.08 [0.801 to 1.45] | 2.67 [2.18 to 3.27] | 0.377 [0.200 to 0.710] | 2.92 [2.33 to 3.65]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.75, 90% CI 2-sided [0.57 to 0.98] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.40, 90% CI 2-sided [0.31 to 0.53] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.13, 90% CI 2-sided [0.08 to 0.22] — GMR is ratio of Experimental Group / Healthy Group

21. Secondary Outcome: Part 1: Fraction of MK-3866 Excretion (Urine) During Each Collection Interval (Fe0-24)
Description: Urine samples were collected at pre-specified intervals and Fe0-24 was assessed. Fe0-24 was obtained by dividing the amount of MK-3866 excreted in each collection interval by the dose. Urine concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Fraction of MK-3866 Excreted
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Healthy Participants (Mild + Moderate RI) | Part 1: Severe Renal Impairment | Part 1: Healthy Participants (Severe RI)
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 9
Fraction of MK-3866 Excreted | 0.485 [0.398 to 0.592] | 0.346 [0.242 to 0.494] | 0.537 [0.445 to 0.648] | 0.173 [0.114 to 0.263] | 0.575 [0.482 to 0.686]
Statistical Analysis 1: Comparison: Part 1: Mild Renal Impairment (RI) vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.90, 90% CI 2-sided [0.74 to 1.11] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 2: Comparison: Part 1: Moderate Renal Impairment vs Part 1: Healthy Participants (Mild + Moderate RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.64, 90% CI 2-sided [0.47 to 0.88] — GMR is ratio of Experimental Group / Healthy Group
Statistical Analysis 3: Comparison: Part 1: Severe Renal Impairment vs Part 1: Healthy Participants (Severe RI); Test type: Other; Geometric Least Squares Mean Ratio (GMR) = 0.30, 90% CI 2-sided [0.21 to 0.43] — GMR is ratio of Experimental Group / Healthy Group

22. Secondary Outcome: Part 2: Total Amount of MK-3866 Excreted Unchanged in the Urine Over the Period of 24 Hours (Ae0-24)
Description: Urine samples were collected at pre-specified intervals and Ae0-24 was assessed. Ae0-24 was obtained by adding the amounts excreted over each collection interval. Urine concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1 of Period 1 and Period 2
Population: All participants who received MK-3866 infusion and provided samples for the outcome. Healthy participants were those who matched gender, and mean age and BMI of the comparator experimental group(s).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 2 | 2 | 8
mg | 4.31 (42.6) | 2.21 (4.4) | 115 (24.9)

23. Secondary Outcome: Part 2: Renal Clearance (CLr) of MK-3866
Description: Urine samples were collected at pre-specified intervals and CLr was assessed. CLr was calculated as AE(t'-t")/AUC(t'-t"), where t'-t" is the longest interval of time during which AE and AUC are both obtained. Urine concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1 of Period 1 and Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 2 | 2 | 8
L/hr | 0.0474 (8.5) | 0.0558 (15.8) | 2.92 (32.1)

24. Secondary Outcome: Part 2: Fraction of MK-3866 Excretion (Urine) During Each Collection Interval (Fe0-24)
Description: Urine samples were collected at pre-specified intervals and Fe0-24 was assessed. Fe0-24 was obtained by dividing the amount of MK-3866 excreted in each collection interval by the dose. Urine concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: Predose and 0-4, 4-8, 8-12, and 12-24 hours after dosing on Day 1 of Period 1 and Period 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fraction of MK-3866 Excreted
Arm/Group | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants (ESRD)
Number analyzed (Participants) | 2 | 2 | 8
Fraction of MK-3866 Excreted | 0.0216 (42.6) | 0.0111 (4.4) | 0.574 (24.9)

25. Secondary Outcome: Part 2: Concentration of MK-3866 in Plasma Entering the Dialyzer Line (Ca)
Description: Plasma samples entering the dialyzer line were collected at pre-specified time points and Ca was assessed. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: All participants who received MK-3866 infusion and provided samples for the outcome. This outcome applied only to ESRD participants receiving HD after infusion of MK-3866 (Part 2, Period 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM
  0.75 hours after dosing | 17.6 (15.6)
  1 hour after dosing | 12.0 (35.8)
  1.5 hours after dosing | 8.67 (33.1)
  2 hours after dosing | 7.25 (10.8)
  2.5 hours after dosing | 5.75 (8.5)
  3 hours after dosing | 4.32 (35.8)
  3.5 hours after dosing | 3.98 (10.3)
  4 hours after dosing | 2.98 (31.8)
  4.5 hours after dosing | 2.57 (31.0)

26. Secondary Outcome: Part 2: Concentration of MK-3866 in Plasma Exiting the Dialyzer Line (Cv)
Description: Plasma samples exiting the dialyzer line were collected at pre-specified time points and Cv was assessed. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM
  0.75 hours after dosing | 8.32 (20.7)
  1 hour after dosing | 7.16 (24.0)
  1.5 hours after dosing | 5.17 (25.1)
  2 hours after dosing | 3.71 (10.5)
  2.5 hours after dosing | 2.92 (11.4)
  3 hours after dosing | 2.69 (21.0)
  3.5 hours after dosing | 2.12 (25.2)
  4 hours after dosing | 2.10 (33.8)
  4.5 hours after dosing | 1.66 (49.4)

27. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of MK-3866 in Plasma Entering the Dialyzer Line During the Dialysis Period (AUCD)
Description: Plasma samples entering the dialyzer line were collected at pre-specified time points and AUCD was assessed. AUCD values were determined from the Ca versus time profile during the HD period, using the 'linear up, log down' calculation method. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM*hr | 29.4 (14.3)

28. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of MK-3866 in Plasma Entering the Dialyzer Line From 0.75 to 4.5 Hours During the Dialysis Period (AUC[0.75-4.5]Ca)
Description: Plasma samples entering the dialyzer line were collected at pre-specified time points and AUC[0.75-4.5]Ca was assessed. AUC[0.75-4.5]Ca values were determined from the Ca versus time profile from 0.75 to 4.5 hours during the HD period, using the 'linear up, log down' calculation method. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM*hr | 23.9 (19.0)

29. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of MK-3866 in Plasma Entering the Dialyzer Line From 0.75 to 4.5 Hours During the Dialysis Period (AUC[0.75-4.5]Cv)
Description: Plasma samples entering the dialyzer line were collected at pre-specified time points and AUC[0.75-4.5]Cv was assessed. AUC[0.75-4.5]Cv values were determined from the Cv versus time profile from 0.75 to 4.5 hours during the HD period, using the 'linear up, log down' calculation method. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µM*hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM*hr | 13.6 (12.2)

30. Secondary Outcome: Part 2: Dialysis Clearance of MK-3866 Based on Plasma (CLD,Plasma)
Description: Plasma dialysis samples were collected at pre-specified time points and CLD was assessed. CLD was calculated as Q x R x (AUC[1-4.5]Ca - AUC[1-4.5]Cv) / AUC[1-4.5]Ca, where Q is the flow rate of blood through the dialyzer, and R is the ratio of blood drug concentration to plasma drug concentration. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
L/hr | 4.81 (201.1)

31. Secondary Outcome: Part 2: Concentration of MK-3866 in Dialysate Samples (CD)
Description: Plasma dialysis samples were collected at pre-specified time points and CD was assessed. Concentrations of MK-3866 were determined using HPLC-MS/MS.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
µM
  0.5 hours after dosing | 1.07 (1.84)
  1 hour after dosing | 3.02 (0.748)
  1.5 hours after dosing | 2.29 (0.153)
  2 hours after dosing | 1.62 (0.142)
  2.5 hours after dosing | 1.30 (0.134)
  3 hours after dosing | 1.08 (0.106)
  3.5 hours after dosing | 0.894 (0.0896)
  4 hours after dosing | 0.695 (0.114)
  4.5 hours after dosing | 0.542 (0.251)

32. Secondary Outcome: Part 2: Amount of MK-3866 Recovered From Each Dialysate Sample (AD)
Description: Plasma dialysis samples were collected at pre-specified time points and AD was assessed. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
mg
  0.5 hours after dosing | 0.946 (8.6)
  1 hour after dosing | 0.736 (31.8)
  1.5 hours after dosing | 0.576 (6.8)
  2 hours after dosing | 0.408 (8.7)
  2.5 hours after dosing | 0.327 (10.7)
  3 hours after dosing | 0.272 (10.3)
  3.5 hours after dosing | 0.224 (10.3)
  4 hours after dosing | 0.173 (17.2)
  4.5 hours after dosing | 0.158 (13.7)

33. Secondary Outcome: Part 2: Rate of Removal of MK-3866 From the Dialysate (rr)
Description: Plasma dialysis samples were collected at pre-specified time points and rr was assessed. rr was calculated as CD x dialysate flow rate. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
mg/hr
  0.5 hours after dosing | 56.7 (8.6)
  1 hour after dosing | 44.2 (31.8)
  1.5 hours after dosing | 34.6 (6.8)
  2 hours after dosing | 24.5 (8.7)
  2.5 hours after dosing | 19.6 (10.7)
  3 hours after dosing | 16.3 (10.3)
  3.5 hours after dosing | 13.5 (10.3)
  4 hours after dosing | 10.4 (17.2)
  4.5 hours after dosing | 9.51 (13.7)

34. Secondary Outcome: Part 2: Cumulative Amount of MK-3866 Recovered From the Dialysate (AD,Total)
Description: Plasma dialysis samples were collected at pre-specified time points and AD,total was assessed. AD,total was obtained by integrating the rr versus time profile over the dialysis session duration, using actual times relative to the start time of dialysis. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
mg | 89.0 (9.3)

35. Secondary Outcome: Part 2: Hemodialysis Clearance of MK-3866 Based on the Dialysate(CLD,Dialysate)
Description: Plasma dialysis samples were collected at pre-specified time points and CLD,dialysate was assessed. CLD,dialysate was calculated as AD.total / AUCD. Concentrations of MK-3866 were determined using HPLC-MS/MS. Method of dispersion used for these data is geometric %CV.
Time Frame: 0.5 (beginning of HD), 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after dosing on Day 1 of Period 2
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD)
Number analyzed (Participants) | 7
L/hr | 6.01 (13.2)

36. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Part 1: up to Day 14 after dosing; Part 2, Period 1: up to Day 14 after dosing (including ≥6 day washout period); Part 2, Period 2: up to Day 14 after dosing
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Healthy Participants: Participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender and mean age and BMI of the comparator groups.
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 10
Participants | 3 | 3 | 1 | 1 | 1 | 1

37. Secondary Outcome: Number of Participants Discontinuing the Study Due to an Adverse Event
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 10
Participants | 0 | 0 | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Part 1: up to Day 14 after dosing; Part 2, Period 1: up to Day 14 after dosing (including ≥6 day washout period); Part 2, Period 2: up to Day 14 after dosing
Description: All participants who received MK-3866 infusion. Healthy participants were those who matched gender, and mean age and BMI of the comparator experimental group(s).
Groups:
- Part 1: Healthy Participants: Participants received a single IV infusion of MK-3886 200 mg over 30 minutes on Day 1. These healthy participants matched the gender, and mean age and BMI of the comparator groups.
Arm/Group | Part 1: Mild Renal Impairment (RI) | Part 1: Moderate Renal Impairment | Part 1: Severe Renal Impairment | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) | Part 1: Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/8 | 1/7 | 0/10
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8 | 1/8 | 0/8 | 0/7 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Mild Renal Impairment (RI) (N=8) | Part 1: Moderate Renal Impairment (N=8) | Part 1: Severe Renal Impairment (N=8) | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) (N=8) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) (N=7) | Part 1: Healthy Participants (N=10)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Mild Renal Impairment (RI) (N=8) | Part 1: Moderate Renal Impairment (N=8) | Part 1: Severe Renal Impairment (N=8) | Part 2, Period 1: ESRD Undergoing HD (Dosed After HD) (N=8) | Part 2, Period 2: ESRD Undergoing HD (Dosed Before HD) (N=7) | Part 1: Healthy Participants (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will provide separate guidance on the criteria for publication of clinical trial data when contacted for permission to publish.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03259087/Prot_SAP_000.pdf